CLINICAL TRIAL: NCT03188653
Title: Evaluating the Effects of Cleansers on the Skin
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left university
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 1705435580
Record Dates: First submitted 2017-05-30; First posted 2017-06-15 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- CeraVe® Eczema Soothing Body Wash (Active Comparator): One of the 7 forearm locations will be selected to receive CeraVe® Eczema Soothing Body Wash one time only.
  Interventions: Other: CeraVe® Eczema Soothing Body Wash
- Cetaphil® RestoraDerm® Eczema Calming Body Wash (Active Comparator): One of the 7 forearm locations will be selected to receive Cetaphil® RestoraDerm® Eczema Calming Body Wash one time only.
  Interventions: Other: Cetaphil® RestoraDerm® Eczema Calming Body Wash
- Dove® Sensitive Skin Body Wash (Active Comparator): One of the 7 forearm locations will be selected to receive Dove® Sensitive Skin Body Wash one time only.
  Interventions: Other: Dove® Sensitive Skin Body Wash
- Eucerin® Skin Calming Body Wash (Active Comparator): One of the 7 forearm locations will be selected to receive Eucerin® Skin Calming Body Wash one time only.
  Interventions: Other: Eucerin® Skin Calming Body Wash
- Aveeno® Skin Relief Body Wash (Active Comparator): One of the 7 forearm locations will be selected to receive Aveeno® Skin Relief Body Wash one time only.
  Interventions: Other: Aveeno® Skin Relief Body Wash
- MooGoo® Milk Wash (Active Comparator): One of the 7 forearm locations will be selected to receive MooGoo® Milk Wash one time only.
  Interventions: Other: MooGoo® Milk Wash
- Free & Clear Liquid Cleanser (Active Comparator): One of the 7 forearm locations will be selected to receive Free & Clear Liquid Cleanser
  Interventions: Other: Free & Clear Liquid Cleanser

INTERVENTIONS:
Other: CeraVe® Eczema Soothing Body Wash — One of the 7 arm locations will be selected to receive CeraVe® Eczema Soothing Body Wash
  Arms: CeraVe® Eczema Soothing Body Wash
Other: Cetaphil® RestoraDerm® Eczema Calming Body Wash — One of the 7 arm locations will be selected to receive Cetaphil® RestoraDerm® Eczema Calming Body Wash
  Arms: Cetaphil® RestoraDerm® Eczema Calming Body Wash
Other: Dove® Sensitive Skin Body Wash — One of the 7 arm locations will be selected to receive Dove® Sensitive Skin Body Wash
  Arms: Dove® Sensitive Skin Body Wash
Other: Eucerin® Skin Calming Body Wash — One of the 7 arm locations will be selected to receive Eucerin® Skin Calming Body Wash
  Arms: Eucerin® Skin Calming Body Wash
Other: Aveeno® Skin Relief Body Wash — One of the 7 arm locations will be selected to receive Aveeno® Skin Relief Body Wash
  Arms: Aveeno® Skin Relief Body Wash
Other: MooGoo® Milk Wash — One of the 7 arm locations will be selected to receive MooGoo® Milk Wash
  Arms: MooGoo® Milk Wash
Other: Free & Clear Liquid Cleanser — One of the 7 arm locations will be selected to receive Free & Clear Liquid Cleanser
  Arms: Free & Clear Liquid Cleanser

SUMMARY:
This will be a single visit study that will take approximately 2 hours. Up to 50 subjects (up to 25 healthy subjects, and up to 25 subjects with AD) from BUMC dermatology clinics will be enrolled in this study and randomized to receive the 7 cleansers on 7 test spots on their upper extremities. One spot will serve as a control and not receive any cleanser. Each spot will be cleansed with the corresponding cleanser for 15 seconds then rinsed off with tap water. Skin barrier will be measured at baseline, immediately after, 30, 60 and 90 minutes after rinse off.

DETAILED DESCRIPTION:
Up to 50 subjects (up to 25 with healthy skin or 25 with atopic dermatitis) meeting the inclusion criteria will be enrolled in this study. A physical exam will be performed to ensure the subjects have healthy skin versus atopic dermatitis. For atopic dermatitis subjects, AD severity will be graded by the EASI score. Site randomization will be performed to determine which cleansers will be used for each of the 8 test sites (one site will be randomized to act as a control and not receive any cleanser). Baseline skin barrier function (TEWL, pH and hydration) will be measured. Then 1ml of each cleansers will be applied to the corresponding test sites, 2ml of tap water will be added, and lathered in a circular motion for 15 seconds. The sites will then be rinsed off with tap water for 15 seconds. Arms will be padded dry. Barrier functions will be measured again immediately after padding dry, and at 30, 60 and 90 minutes after.

ELIGIBILITY:
Inclusion Criteria:

Male and female, at least 18 years of age Subject must be able to comprehend and read the English language. Healthy skin without concurrent atopic dermatitis or diagnosed with atopic dermatitis by a dermatologist

Exclusion Criteria:

Subjects who do not fit the inclusion criteria. Subjects unable to or unwilling to comply with the study procedures Concurrently have other inflammatory skin conditions. Prior known allergy to any components to of the cleansers tested A subject who, in the opinion of the investigator, will be uncooperative or unable to comply with study procedures.

Subject unable to speak or read the English language, since all consents and instructions will be provided in English.

Those that are prisoners or cognitively impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Skin barrier function | 2 hours
  Transepidermal water loss (TEWL) will be measured using hand-held, noninvasive skin barrier measuring device (VapoMeter).

SECONDARY OUTCOMES:
Skin barrier function | 2 hours
  Stratum corneum hydration status will be measured using hand-held, noninvasive skin barrier measuring device (MoistureMeterSC).
Skin pH | 2 hours
  Skin pH will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona - Banner University Medicine Dermatology, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No